CLINICAL TRIAL: NCT06049277
Title: Effects of Mulligan Technique Versus McKenzie Extension Exercise With Manual Traction in Patients With Chronic Unilateral Radicular Low Back Pain
Brief Title: Mulligan Technique Versus McKenzie Extension Exercise Chronic Unilateral Radicular Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0133 Maira
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Range of Motion; Manual Therapy; Pain; Mobilization
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan techniques with manual traction (Experimental): Mulligan techniques with manual traction
  Interventions: Other: Mulligan techniques with manual traction
- McKenzie extension exercises with manual traction (Active Comparator): McKenzie extension exercises with manual traction
  Interventions: Other: McKenzie extension exercises with manual traction

INTERVENTIONS:
Other: Mulligan techniques with manual traction — group A will be treated with Mulligan techniques with manual traction.16 patients in group A will be treated with Mulligan Techniques SNAGS in sitting, standing and prone position by applying Antero cranial glide in the direction of treatment plane over the spinous or transverse process and Spinal mobilization with leg movement at 6 to 8 repetitions per sessions and spinal mobilization with leg movement will be performed in side lying, patient facing the physiotherapist while the leg movement may assisted by another person (Physiotherapist/assistant). Sustained transverse glide is given on the desired spinous process with 10 repetitions of offending movement in first session while 10 reps in each of 3 sets in further sessions.
  Arms: Mulligan techniques with manual traction
Other: McKenzie extension exercises with manual traction — group B will be treated McKenzie extension exercises with manual traction.16 patients in group B will be treated with McKenzie active EEP in prone position with repeated movements along with standard protocols. McKenzie Extension Exercises performed actively in prone position. Extension exercises performed in three stages, initially patient instructed to be just lift the neck and look on front at the eye level, then progressed next and weight bearing on the elbow by lifting up the shoulder and then moved on third and final steps in which complete trunk extension is performed and weight bearing is on the hands.
  Arms: McKenzie extension exercises with manual traction

SUMMARY:
This project will be a Randomized clinical trial conducted to determine effects of Mulligan technique versus McKenzie extension exercise with manual traction in patients with chronic unilateral radicular low back pain. Sample will be collected through non-probability convenient sampling, following eligibility criteria from Rehab Care and Jinnah Hospital Lahore. Eligibility criteria will be both gender and age range 28-50 years, clinically diagnosed patient with Lumbar radiculopathy after exclusion of the patients with Fracture, Trauma, Inflammatory disorder, acute disc bulge, Lumbar instability. Participants will be randomly allocated in two groups via sealed envelope method, baseline assessment will be done, Group A participants will be given baseline treatment along with Mulligan techniques, Group B participants will be given baseline treatment along with McKenzie protocol. Pre and post intervention assessment will be done via, Numeric pain rating scale(NPRS), Oswestry Disability Scale (ODI) and lumber Range of Motion, 2 sessions per week will be given for 4 weeks, data will be analyzed by using SPSS version 29.

DETAILED DESCRIPTION:
Chronic mechanical low back pain is common among different age groups and genders. Different manual therapy techniques combined with exercise therapy and electrotherapy modalities play an important role in its management. Our objective was to compare the effects of McKenzie extension exercises program versus Mulligan Techniques for chronic unilateral radicular low back pain. The primary objective of my study is to evaluate the outcome of Mulligan technique versus McKenzie extension exercise with manual traction in patients with chronic unilateral radicular low back pain in terms of pain reduction and ROM.

A randomized control trial will be conducted at Rehab Care and Jinnah Hospital Lahore, from 1st June - 31st January 2024. Both genders and age range 28-50 years clinically diagnosed patient with Lumbar radiculopathy will be included. The patients with Fracture, Trauma, Inflammatory disorder, acute disc bulge, Lumbar instability will be excluded. Subjects will be divided into two equal groups through a computer-generated random number. Sixteen patients in group A will be treated with Mulligan techniques and Sixteen patients in group B with McKenzie for four weeks at two session per week and single session per day. Visual Analogue Scale, Oswestry Disability Scale and lumbar Range of Motion will be used as an assessment tool and were measured at baseline and at the completion 4 weeks intervention. The data will be entered and analyzed with SPSS to draw the statistical and clinical significance of both interventions. Results will be presented as mean and standard deviation for numerical variables like Visual Analogue Scale, Oswestry Disability Scale and lumber Range of Motion. Analysis will be done by statistical package for social sciences SPSS 29

ELIGIBILITY:
Inclusion Criteria:

* Age range 28-50 years
* Patients of both gender
* Clinically diagnosed patient with Lumbar radiculopathy

Exclusion Criteria:

* Subject with chronic radicular low back pain with the history of spinal surgery
* Patients who have recently received corticosteroids
* Diagnosed cases of osteoporosis
* History of recent Fracture
* Lumber instability
* Trauma
* Inflammatory disorders
* Acute disc bulge

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
NPRS | 4th Week
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain.
Oswestry Disability Scale (ODI) | 4th Week
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools.
Range of Motion | 4th Week
  Assessment of range of motion (ROM) of the lumbar spine is an important part lumbar spine examination. Range of motion will be measured with inclinometer. Aberrant spinal motion is associated with faulty spinal mechanics. Motion of the lumbar spine will be assessed in all planes including flexion, extension, side bending, and rotation. Variables affect lumbar range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, Principal Investigator — Riphah International University, Lahore, Pakistan; Maira Saeed, Principal Investigator — Riphah International University, Lahore, Pakistan
Locations (1):
- Jinnah Hospital Lahore, Rehab Care, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buran Cirak Y, Yurdaisik I, Elbasi ND, Tutuneken YE, Koce K, Cinar B. Effect of Sustained Natural Apophyseal Glides on Stiffness of Lumbar Stabilizer Muscles in Patients With Nonspecific Low Back Pain: Randomized Controlled Trial. J Manipulative Physiol Ther. 2021 Jul-Aug;44(6):445-454. doi: 10.1016/j.jmpt.2021.06.005. Epub 2021 Aug 26. PMID 34456042
- [Background] Tul Ain SQ, Shakil Ur Rehman S, Maryam M, Kiani SK. Effects of Sustained Natural Apophyseal Glides with and without thoracic posture correction techniques on mechanical back pain: a randomized control trial. J Pak Med Assoc. 2019 Nov;69(11):1584-1587. doi: 10.5455/JPMA.274875.. PMID 31740859
- [Background] Waqqar S, Shakil-Ur-Rehman S, Ahmad S. McKenzie treatment versus mulligan sustained natural apophyseal glides for chronic mechanical low back pain. Pak J Med Sci. 2016 Mar-Apr;32(2):476-9. doi: 10.12669/pjms.322.9127. PMID 27182265
- [Background] Cuesta-Vargas A, Farasyn A, Gabel CP, Luciano JV. The mechanical and inflammatory low back pain (MIL) index: development and validation. BMC Musculoskelet Disord. 2014 Jan 9;15:12. doi: 10.1186/1471-2474-15-12. PMID 24405779
- [Background] O'Sullivan PB, Phyty GD, Twomey LT, Allison GT. Evaluation of specific stabilizing exercise in the treatment of chronic low back pain with radiologic diagnosis of spondylolysis or spondylolisthesis. Spine (Phila Pa 1976). 1997 Dec 15;22(24):2959-67. doi: 10.1097/00007632-199712150-00020. PMID 9431633
- [Background] Chitale N Jr, Patil DS, Phansopkar P, Joshi A. A Review on Treatment Approaches for Chronic Low Back Pain via Mulligans Movement With Mobilization and Physical Therapy. Cureus. 2022 Aug 18;14(8):e28127. doi: 10.7759/cureus.28127. eCollection 2022 Aug. PMID 36134056
- [Background] Salik S RS, Hayaat R, Manzoor S, Malik AU, Maqbool S. Comparison of Mulligan sustained natural apophyseal glides verses Mckenzie extension exercises on disability and functional outcomes in patients with acute nonspecific low back pain. PJMHS. 2022;16(10):1:5.
- [Background] May S, Donelson R. Evidence-informed management of chronic low back pain with the McKenzie method. Spine J. 2008 Jan-Feb;8(1):134-41. doi: 10.1016/j.spinee.2007.10.017. PMID 18164461
- [Background] Almeida MO, Narciso Garcia A, Menezes Costa LC, van Tulder MW, Lin CC, Machado LA. The McKenzie method for (sub)acute non-specific low back pain. Cochrane Database Syst Rev. 2023 Apr 5;4(4):CD009711. doi: 10.1002/14651858.CD009711.pub2. PMID 37017272